CLINICAL TRIAL: NCT02676102
Title: Community Based Research to Improve Organ Donor Registration Among Black Men - Aim 2 Randomized Trial Comparing Tailored Versus Targeted Videos.
Brief Title: RCT Comparing Tailored Versus Targeted Organ Donation Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-02109
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Organ Transplants
Keywords: barber shops; organ transplant; transplants; organ donor registration
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Participant will watch an educational video produced in partnership with the community of black men including customers, employers and owners of BOBs.
  Interventions: Behavioral: Control Group
- Targeted Intervention (Active Comparator): Participants will watch an educational video produced in partnership with the community of black men including customers, employees, and owners of BOBs. Video production was informed by entertainment education models and produced with experts including an Academy Award winning filmmaker.
  Interventions: Behavioral: Targeted Intervention
- Tailored Intervention (Active Comparator): Participants will watch videos with content individualized to participant's pre-intervention ODBI scores representing their organ donation beliefs
  Interventions: Behavioral: Tailored Intervention

INTERVENTIONS:
Behavioral: Control Group — Generic Video about organ donation
  Arms: Control Group
Behavioral: Targeted Intervention — an educational video produced in partnership with the community of black men including customers, employees, and owners of BOBs. Video production was informed by entertainment education models and produced with experts including an Academy Award winning filmmaker.
  Arms: Targeted Intervention
Behavioral: Tailored Intervention — Videos with content individualized to participant's pre-intervention Organ Donation Belief Index (ODBI).
  Arms: Tailored Intervention

SUMMARY:
The primary purpose of this 3-phase mixed methods design study is to investigate how presenting content at varying levels of audience specificity (generic, targeted, and tailored) influences organ donor registration behavior among black men using video-based educational programming produced and distributed in partnership with our network of Black Owned Barbershops (BOBs). Investigators have completed a development phase using digital video interviewing to both derive and provide culturally specific content for the videos. This phase of this investigation is a 3 arm randomized control trial (RCT) phase, in which customers will be randomized to receive the generic, targeted, or tailored video programming delivered with iPads, after which an immediate organ donation opportunity will be offered through registration online or with a mailed in application. The final phase of this investigation will be a failure analysis whereby we will interview a subset of participants who registered or failed to register one month after their educational session to ascertain how the programming impacted their decision (Aim 3 - the subject of a future IRB application).

ELIGIBILITY:
Inclusion Criteria:

* Black men who visit BOBs
* Participants whose primary language is English
* Participants who reside locally in NYC for at least four weeks (28 days) in a year

Exclusion Criteria:

* Women are excluded from this study, as it is focused on black men who visit BOBs, who are among the most in need for transplants, and least likely to register as organ donors.
* Women are excluded from this study, as it is focused on black men who visit BOBs, who are among the most in need for transplants, and least likely to register as organ donors.
* Persons not self-reporting being a black male are excluded. Including other minority groups would preclude conducting this research given its budget and time constraints.
* Children under 18 years old are excluded from this research.
* Persons who are visually impaired and are unable to watch the videos.
* Persons who are hearing impaired and are unable to hear the audio on the videos.
* Persons who self report to be registered in the New York State Organ Donor Registry.
* Persons who are cognitively impaired and thus are unable to provide consent to register for organ donation by signing the New York State Organ Donor Registry application.
* Persons who previously are enrolled in this randomized controlled trial. Women are excluded from this study, as it is focused on black men who visit BOBs, who are among the most in need for transplants, and least likely to register as organ donors.
* Persons not self-reporting being a black male are excluded. Including other minority groups would preclude conducting this research given its budget and time constraints.
* Children under 18 years old are excluded from this research.
* Persons who are visually impaired and are unable to watch the videos.
* Persons who are hearing impaired and are unable to hear the audio on the videos.
* Persons who self report to be registered in the New York State Organ Donor Registry.
* Persons who are cognitively impaired and thus are unable to provide consent to register for organ donation by signing the New York State Organ Donor Registry application.
* Persons who previously are enrolled in this randomized controlled trial. Persons not self-reporting being a black male are excluded. Including other minority groups would preclude conducting this research given its budget and time constraints.
* Children under 18 years old are excluded from this research.
* Persons who are visually impaired and are unable to watch the videos.
* Persons who are hearing impaired and are unable to hear the audio on the videos.
* Persons who self report to be registered in the New York State Organ Donor Registry.
* Persons who are cognitively impaired and thus are unable to provide consent to register for organ donation by signing the New York State Organ Donor Registry application.
* Persons who previously are enrolled in this randomized controlled trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1440 (Actual)
Dates: Start 2015-02; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of Immediate Registrations | 1 Day
  Enrollment number in the the NY State Organ Donor Registry

SECONDARY OUTCOMES:
Number of Confirmed Registrations | 1 Day
  Post Intervention NY State Department of Health aggregate data by video group
Number of participants that viewed "How To Register" Video | 1 Day
  Post Intervention research assistant assisted / observed
Accepted Information Score | 1 Day
  Post Intervention RA assisted / observed
Organ Donation Beliefs (ODBI) Survey Score | 1 Day
  Pre-Intervention iPad Survey

OTHER OUTCOMES:
Participant Demographics | 1 Day
  Age, education, religion, sex, race

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wall, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States